CLINICAL TRIAL: NCT04360551
Title: Randomized, Double-Blind, Placebo-Controlled Pilot Clinical Trial of the Safety and Efficacy of Telmisartan for the Mitigation of Pulmonary and Cardiac Complications in COVID-19 Patients
Brief Title: Pilot Clinical Trial of the Safety and Efficacy of Telmisartan for the Mitigation of Pulmonary and Cardiac Complications in COVID-19 Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Decrease in COVID-19 cases locally
Sponsor: University of Hawaii (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H051; U54MD007601-34S3 (NIH)
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Telmisartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Placebo controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Telmisartan (Experimental): Telmisartan 40 mg po daily x 21 days
  Interventions: Drug: Telmisartan 40mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Telmisartan 40mg — Angiotensin Receptor Blocker (ARB)
  Arms: Telmisartan
Drug: Placebo — Placebo once daily
  Arms: Placebo

SUMMARY:
This study will enroll 40 symptomatic outpatients tested positive for Coronavirus 2019 (COVID-19). Patients to be randomized 1:1 to Telmisartan (40 mg) vs placebo to be administered orally once daily x 21 days. Daily, the study patients will be asked to keep a record of the severity of their fever, dyspnea and fatigue and take their blood pressure (BP) and temperature. Study visits to occur on day 1 (entry), day 4, day 10 and day 21. Oro-pharyngeal swabs, and approximately 25 cc of blood will be collected at each study visit for safety labs and for the evaluation of the renin-angiotensin system (RAS) system and for various blood biomarkers of inflammation, coagulation and fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent prior to initiation of any study procedures.
* Understands and agrees to comply with planned study procedures including self testing of blood pressure daily
* Male or non-pregnant female adult ≥18 years of age at time of enrolment.
* Has laboratory-confirmed severe acute respiratory syndrome corona virus 2 (SARS-CoV-2) infection as determined by FDA-approved commercial or public health assay in any specimen collected ideally < 72 hours prior to randomization. Exceptions to the <72 hr inclusion criteria may be made at the discretion of the investigator.
* Positive for COVID-19 symptoms: fever defined as a temperature of >100.4 on study screening or self-report of daily fever at home OR shortness of breath of any degree OR fatigue causing greater than minimal interference with usual social & functional activities
* Women of childbearing potential must agree to use at least one primary form of contraception for the duration of the study
* Able to easily swallow pills

Exclusion Criteria:

* Immediate need for hospitalization on screening
* Systolic blood pressure less than 100 mmHg
* Self-reported presence of chronic kidney disease or requiring dialysis
* Self-reported history of liver failure or untreated hepatitis B or C
* Pregnancy or breast feeding
* Allergy to the study medication
* Current use of angiotensin receptor blocker (ARB) or angiotensin converting enzyme (ACE) Inhibitor medications. Other blood pressure medications will be permitted in the systolic BP is higher than 90 mmHg
* Prior reaction or intolerance to ARB or ACE Inhibitor
* Use of aliskiren in patients with diabetes
* Current use of and on-going need for lithium, digoxin, potassium sparing diuretics such as spironolactone
* Current use of and need for potassium supplements
* Current or past participation in a research study within 12 weeks prior to the Screening Visit unless cleared by Study Team
* Inability to drive safely for study visits
* Subjects, who, in the opinion of the investigator, are unable to comply with the protocol evaluation, or for whom study participation may not be advisable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia M Shikuma, MD, Principal Investigator — University of Hawaii at Manoa John A Burns School of Medicine
Locations (1):
- University of Hawaii - Manoa, John A Burns School of Medicine UH Clinics at Kakaako, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was advertised generally via physicians and clinics connected with our research center as well as via our medical school's community relations outreach office. Because of the communicable nature of acute COVID-19 infection, the participants were screened, enrolled and underwent their study visits under a portable tent just outside our research clinic on the grounds of the medical school.
Pre-assignment Details: No pre-assignment events.
Period: Overall Study
Arm/Group | Telmisartan | Placebo
Started | 12 | 12
Completed | 11 | 12
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telmisartan | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years]
  mean age | 35.83 (12.445) | 35.83 (11.991) | 35.83 (11.952)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 8 | 4 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian Asian | 2 | 4 | 6
  Native Hawaiian/Pacific Islander | 3 | 3 | 6
  Black | 0 | 0 | 0
  White | 4 | 3 | 7
  More than One Race | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
Clinical Status [Median (Inter-Quartile Range); unit: units on a scale] — Clinical status of the participant at BASELINE based on a 7-point Clinical Status ordinal scale adapted from the WHO MASTER PROTOCOL for the Treatment of COVID-19 in Hospitalized Patients modified to allow inclusion of a symptom scale for non-hospitalized patients from grade 1 to 4 for fever, dyspnea and fatigue to further define individuals within WHO scale '2' defined as 'not hospitalized, limited on activities'.
  units on a scale | 2.125 [2.00 to 2.25] | 2.00 [2.00 to 2.25] | 2.00 [2.00 to 2.25]

OUTCOME MEASURES:

1. Primary Outcome: Maximum Clinical Severity of Disease Since Entry
Description: We utilized the World Health Organization (WHO) COVID-19 7-point ordinal scale: 1 (not hospitalized, no limitations on activities), 2 (not hospitalized limitation on activities); 3 (hospitalized, not requiring oxygen); 4 (hospitalized and requiring oxygen); 5 (hospitalized, on non-invasive ventilation or high flow oxygen devices); 6 (hospitalized, on invasive mechanical ventilation or ECMO) and 7 (death).
  A symptom scale was devised to allow 'fine tuning' within the 2.0 WHO category of 'not hospitalized but limitation on activities' based on severity (no symptoms, mild, moderate, moderately severe and severe symptoms) of fever, breathing and fatigue severity scale (0 to 4 points for each factor allowing a max score of 12). A WHO scale within the '2' category was then 'fine tuned' as follows: 2.0 (</=3 symptom points), 2.25 (4-6 symptom points), 2.5 (7-9 symptom points), and 2.75 (10-12 symptom points).
Time Frame: maximum clinical severity of disease post entry evaluated over the 21 day clinical study
Population: Participants with acute COVID infection and symptoms
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Telmisartan | Placebo
Number analyzed (Participants) | 12 | 12
score on a scale | 2.00 [2.00 to 2.00] | 2.000 [2.00 to 2.25]
Statistical Analysis 1: Comparison: Telmisartan vs Placebo; Test type: Superiority; p = 0.244, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number of Adverse Events
Description: Number of adverse events grade 2 and above utilizing the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.0, November 2014
Time Frame: Through study completion at day 21 of study
Population: All participants entered into the study
Measure: Number; unit: adverse events
Arm/Group | Telmisartan | Placebo
Number analyzed (Participants) | 12 | 12
adverse events
  headache | 1 | 1
  nasal congestion | 1 | 1
  shortness of breath | 0 | 1
  nausea | 1 | 0
  diarrhea | 1 | 0
  chest discomfort | 1 | 0
Statistical Analysis 1: Comparison: Telmisartan vs Placebo; Test type: Superiority; p > 0.5, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: During the 21 days of the study.
Description: Same definition of adverse events and serious adverse events were used.
Groups:
- Telmisartan Arm: Randomized to receive Telmisartan
- Placebo Arm: Randomized to placebo
Arm/Group | Telmisartan Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telmisartan Arm (N=12) | Placebo Arm (N=12)
headache (Nervous system disorders) | 1 (1) | 1 (1)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
chest discomfort (Cardiac disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The number of individuals involved in the study was extremely small. The study was terminated early because the number of infections in the community substantially decreased.

As an outpatient study, the study only involved individuals with mild to moderate COVID-19 infection, as those severely ill with acute COVID-19 infections may have been hospitalized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/51/NCT04360551/Prot_SAP_000.pdf